CLINICAL TRIAL: NCT02411903
Title: The Dynamic Effect of Non-cytochrome P450 Isoenzyme 3A4（CYP3A4）-Metabolized and Cytochrome P450 Isoenzyme 3A4（CYP3A4）-Metabolized Statins on Clopidogrel Resistance in Patients With Cerebral Infarction
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: The Third Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Bo Rong Zhou, chief physicians, The Third Affiliated Hospital of Guangzhou Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H0906
Record Dates: First submitted 2015-03-17; First posted 2015-04-08 (Estimated); Last update posted 2015-06-16 (Estimated); Status verified 2015-04

CONDITIONS: Cerebral Infarction; Clopidogrel,Poor Metabolism of (Disorder)
Keywords: Clopidogrel-drug interactions
MeSH Terms: conditions — Cerebral Infarction | interventions — Atorvastatin; Clopidogrel; Rosuvastatin Calcium

ARMS (2):
- atorvastatin and Clopidogrel (Active Comparator): 80 patients will be taking atorvastatin 40mg/d plus clopidogrel 75mg/d for 9 months。
  Interventions: Drug: atorvastatin and clopidogrel
- rosuvastatin and Clopidogrel (Experimental): 80 patients will be taking rosuvastatin 20mg/d plus clopidogrel 75mg/d for 9 months。
  Interventions: Drug: rosuvastatin and clopidogrel

INTERVENTIONS:
Drug: atorvastatin and clopidogrel — Dose: atorvastatin 40mg/d plus clopidogrel 75mg/d for 9 months.
  Arms: atorvastatin and Clopidogrel
Drug: rosuvastatin and clopidogrel — Dose: rosuvastatin 20mg/d plus clopidogrel 75mg/d for 9 months.
  Arms: rosuvastatin and Clopidogrel

SUMMARY:
The investigators team had found that the presence of dynamic changes of Clopidogrel resistance are not associated with genetic factors. Currently, study on moderate doses of statins and dynamic Clopidogrel resistance has not been reported, therefore this study will observe 160 cases of open prospective secondary prevention in patients with cerebral infarction. Excluded: those patients occurs Clopidogrel resistance because of slow metabolism caused by cytochrome P450 isoenzyme 2C19（CYP2C19, and then observed the impact of the cytochrome P450 isoenzyme 3A4 （CYP3A4）-metabolized and non-cytochrome P450 isoenzyme 3A4 （CYP3A4）-metabolized statins dynamically on Clopidogrel resistance in the next 9 months, adverse events will be recorded, the metabolite of clopidogrel（H4 ）and the polymorphism of cytochrome P450 isoenzyme 2C19 （CYP2C19）/cytochrome P450 isoenzyme 3A4 （CYP3A4）/ cytochrome P450 isoenzyme 2C9（CYP2C9）will be detected. Expected Result: the patients use the cytochrome P450 isoenzyme 3A4（CYP3A4）-metabolized statins will result in dynamic Clopidogrel resistance easily ,H4 levels will decline, and Clopidogrel resistance is not related to the polymorphism of cytochrome P450 isoenzyme 3A4 （CYP3A4）.

ELIGIBILITY:
Inclusion Criteria:

* The patient must have signed an informed consent document indicating that they understand the purpose of and procedures required for the study and are willing to participate in the study.
* Age <85 years and >45 years ,Male or female.
* The patient have been Cerebral infarction for one month.
* national institutes of health stroke scale（NIHSS）score ≤23 points.
* Blood Platelet count greater than 150×10^9／L,and Less than 500×10^9／L.
* The patient never do not taking aspirin 、dipyridamole、clopidogrel,or the patient had been taken these anti-platelet drugs but has been discontinued for two weeks at least.
* The patient never do not taking Statins or the patient have been stop taking statins 2 weeks for two weeks.

Exclusion Criteria:

* Allergic constitution , or allergic to the composition of the drugs in this study.
* national institutes of health stroke scale（NIHSS） score >23 points.
* Atrial fibrillation and other cardiogenic cerebral embolism.
* Patients who were undergone surgery and trauma (including fractures) within the past three month.
* Patients with known dysfunction of vital organs or suffered from Serious cardiovascular disease ，or coagulation disorders.
* The patient took Proton pump inhibitors recently.
* The history of data collection and the follow-up process can not be saved.

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2015-03; Primary Completion 2016-07 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
incidence of clopidogrel resistance | For nine months
  Definition of clopidogrel resistance is the absolute change of 5 microliter adenosine diphosphate(ADP) induced PAR≤10% as compared to baseline. So, incidence of clopidogrel resistance= (PAR at monitor point - PAR at baseline) / PAR at baseline×100 %≤10 %。 Measures of PAR: PAR is measured by Light transmittance aggregometry (LTA) and according to the standard of Rev。

REFERENCES:
- [Result] Sugunaraj JP, Palaniswamy C, Selvaraj DR, Chaitanya Arudra SK, Sukhija R. Clopidogrel resistance. Am J Ther. 2010 Mar-Apr;17(2):210-5. doi: 10.1097/MJT.0b013e3181bdc3e4. PMID 19829090
- [Result] Nguyen TA, Diodati JG, Pharand C. Resistance to clopidogrel: a review of the evidence. J Am Coll Cardiol. 2005 Apr 19;45(8):1157-64. doi: 10.1016/j.jacc.2005.01.034. PMID 15837243
- [Result] Lev EI, Patel RT, Maresh KJ, Guthikonda S, Granada J, DeLao T, Bray PF, Kleiman NS. Aspirin and clopidogrel drug response in patients undergoing percutaneous coronary intervention: the role of dual drug resistance. J Am Coll Cardiol. 2006 Jan 3;47(1):27-33. doi: 10.1016/j.jacc.2005.08.058. Epub 2005 Dec 9. PMID 16386660